CLINICAL TRIAL: NCT03715829
Title: A PHASE 2B RANDOMIZED, DOUBLE-BLIND, PLACEBO-CONTROLLED, MULTICENTER, DOSE-RANGING STUDY TO EVALUATE THE EFFICACY AND SAFETY PROFILE OF PF-06651600 WITH A PARTIALLY BLINDED EXTENSION PERIOD TO EVALUATE THE EFFICACY AND SAFETY OF PF-06651600 AND PF-06700841 IN SUBJECTS WITH ACTIVE NON-SEGMENTAL VITILIGO
Brief Title: A Phase 2b Study To Evaluate The Efficacy And Safety Profile Of PF-06651600 And PF-06700841 In Active Non-segmental Vitiligo Subjects
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Pfizer (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: B7981019; 2018-001271-20 (EudraCT Number)
Record Dates: First submitted 2018-10-19; First posted 2018-10-23 (Actual); Results first posted 2022-03-25 (Actual); Last update posted 2022-03-25 (Actual); Status verified 2022-03

CONDITIONS: Active Non-segmental Vitiligo
MeSH Terms: interventions — PF-06651600; PF-06700841

STUDY DESIGN:
Intervention Model Description: Dose ranging period is a parallel design. Extension period is a sequential design.
Who Masked: Participant, Investigator, Outcomes Assessor
Masking Description: Dose ranging period is blinded. The partially blinded extension period includes open arms and blinded arms.
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (12):
- Cohort 1 (Experimental): Induction dose 1 given once a day(QD) for 4 weeks followed by maintenance dose A given QD for 20 weeks
  Interventions: Drug: PF-06651600
- Cohort 2 (Experimental): Induction dose 2 given QD for 4 weeks followed by maintenance dose A given QD for 20 weeks
  Interventions: Drug: PF-06651600
- Cohort 3 (Experimental): Maintenance dose A given QD for 24 weeks
  Interventions: Drug: PF-06651600
- Cohort 4 (Experimental): Maintenance dose B given QD for 24 weeks
  Interventions: Drug: PF-06651600
- Cohort 5 (Experimental): Maintenance dose C given QD for 24 weeks
  Interventions: Drug: PF-06651600
- Cohort 6 (Placebo Comparator): Placebo given QD for 24 weeks
  Interventions: Drug: placebo
- Extension Cohort 1 (Experimental): 4 week drug holiday (no drug given) followed by PF-06700841 oral tablet QD for 20 weeks
  Interventions: Drug: PF06700841
- Extension Cohort 2 (Experimental): Induction dose 1 given QD for 4 weeks followed by maintenance dose A given QD for 20 weeks in conjunction with narrow band UVB phototherapy
  Interventions: Drug: PF-06651600; Device: narrow-band UVB phototherapy
- Extension Cohort 3 (Experimental): Induction dose 1 given QD for 4 weeks followed by maintenance dose A given QD for 20 weeks
  Interventions: Drug: PF-06651600
- Extension Cohort 4 (Experimental): Maintenance dose A given QD for 24 weeks
  Interventions: Drug: PF-06651600
- Extension Cohort 5 (Experimental): Maintenance dose B given QD for 24 weeks
  Interventions: Drug: PF-06651600
- Extension Cohort 6 (No Intervention): Observation period for 24 weeks

INTERVENTIONS:
Drug: PF-06651600 — Induction dose 1. Oral tablet taken QD
  Arms: Cohort 1; Extension Cohort 2; Extension Cohort 3
Drug: PF-06651600 — Induction dose 2. Oral tablet taken QD
  Arms: Cohort 2
Drug: PF-06651600 — Maintenance dose A. Oral tablet taken QD
  Arms: Cohort 1; Cohort 2; Cohort 3; Extension Cohort 2; Extension Cohort 3; Extension Cohort 4
Drug: PF-06651600 — Maintenance Dose B. Oral tablet taken QD
  Arms: Cohort 4; Extension Cohort 5
Drug: PF-06651600 — Maintenance Dose C. Oral tablet taken QD
  Arms: Cohort 5
Drug: placebo — placebo
  Arms: Cohort 6
Drug: PF06700841 — Oral tablet taken QD
  Arms: Extension Cohort 1
Device: narrow-band UVB phototherapy — Phototherapy will be combined with PF-06651600
  Arms: Extension Cohort 2

SUMMARY:
This is a Phase 2b, randomized, double blind, parallel group, multicenter study with an extension period. The study will have a maximum duration of approximately 60 weeks. This includes an up to 4 weeks Screening Period, a 24 week dose ranging period, an up to 24 week extension period and a 8 week Follow up Period.

ELIGIBILITY:
Inclusion Criteria:

* Male or female subjects between 18-65 years of age, inclusive, at time of informed consent.
* Must have moderate to severe active non-segmental vitiligo.

Exclusion Criteria:

* History of human immunodeficiency virus (HIV) or positive HIV serology at screening,
* Infected with hepatitis B or hepatitis C viruses.
* Have evidence of active or latent or inadequately treated infection with Mycobacterium tuberculosis (TB)

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 366 (Actual)
Dates: Start 2018-11-26 (Actual); Primary Completion 2021-02-05 (Actual); Study Completion 2021-02-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (90):
- United States (40):
  - Marvel Research, LLC, Huntington Beach, California
  - University of California, Irvine, Dermatology Clinical Research Center, Irvine, California
  - Vitiligo and Pigmentation Institute Of Southern California, Los Angeles, California
  - Dermatology Specialist, Inc., Murrieta, California
  - Dermatology Specialists, Inc., Oceanside, California
  - UC Davis Health, Sacramento, California
  - Brookside Dermatology Associates, Bridgeport, Connecticut
  - New England Research Associates, LLC, Bridgeport, Connecticut
  - New Horizon Research Center, Miami, Florida
  - Park Avenue Dermatology, Orange Park, Florida
  - ForCare Clinical Research, Tampa, Florida
  - Advanced Skin and MOHS Surgery Center, c/o TrialSpark, Inc., Chicago, Illinois
  - Chevy Chase Dermatology Center (TrialSpark, Inc.), Chevy Chase, Maryland
  - TrialSpark - Samantha Toerge, MD, Chevy Chase, Maryland
  - TrialSpark - Ronald Shore, MD, Rockville, Maryland
  - Tobias & Battite, Inc., Boston, Massachusetts
  - Tufts Medical Center, Boston, Massachusetts
  - UMass Memorial Medical Center, Hahnemann Campus, Worcester, Massachusetts
  - Investigational Drug Service Pharmacy, Worcester, Massachusetts
  - UMass Memorial Medical Center Ear Nose and Throat, Worcester, Massachusetts
  - University of Massachusetts Medical School, Worcester, Massachusetts
  - Henry Ford Hospital Department of Dermatology, Detroit, Michigan
  - University of Minnesota Department of Dermatology, Minneapolis, Minnesota
  - The Dermatology Group, P.C., Verona, New Jersey
  - Icahn School of Medicine at Mount Sinai, New York, New York
  - Upper West Side Dermatology c/o TrialSpark, Inc, New York, New York
  - MDCS: Medical Dermatology & Cosmetic Surgery (TrialSpark, Inc.), New York, New York
  - South Nassau Dermatology, Oceanside, New York
  - TrialSpark, Inc. - Russell W. Cohen, MD, Oceanside, New York
  - PMG Research of Wilmington, LLC, Wilmington, North Carolina
  - Remington-Davis, Inc. Clinical Research, Columbus, Ohio
  - ForeFront Dermatology, Columbus, Ohio
  - Vital Prospects Clinical Research Institute, PC, Tulsa, Oklahoma
  - University Physicians Group, Austin, Texas
  - University of Texas Southwestern Medical Center, Dallas, Texas
  - Pickens Academic Tower, Houston, Texas
  - The University of Texas Health Science Center at Houston, Houston, Texas
  - The University of Texas MD Anderson Cancer Center, Houston, Texas
  - Virginia Clinical Research, Inc, Norfolk, Virginia
  - Tamjidi Skin Institute (TrialSpark, Inc.), Vienna, Virginia
- Australia (6):
  - The Skin Hospital, Darlinghurst, New South Wales
  - Premier Specialists Pty Ltd, Kogarah, New South Wales
  - Veracity Clinical Research Pty Ltd, Woolloongabba, Queensland
  - Skin Health Institute, Carlton, Victoria
  - Sinclair Dermatology, East Melbourne, Victoria
  - The Royal Melbourne Hospital, Parkville, Victoria
- Belgium (3):
  - Hôpital Erasme Dermatology, Brussels
  - UZ Brussel - Dermatology, Brussels
  - UZ Gent - Dermatology, Ghent
- Canada (16):
  - Dr. Chih-ho Hong Medical Inc., Surrey, British Columbia
  - Enverus Medical Research, Surrey, British Columbia
  - University of British Columbia, Vancouver, British Columbia
  - Wiseman Dermatology Research Inc., Winnipeg, Manitoba
  - CCA Medical Research, Ajax, Ontario
  - Guenther Research Inc., London, Ontario
  - Lynderm Research Inc., Markham, Ontario
  - DermEdge Research, Mississauga, Ontario
  - North York Research Inc., North York, Ontario
  - The Centre for Clinical Trials, Oakville, Ontario
  - The Centre for Dermatology, Richmond Hill, Ontario
  - K.Papp Clinical Research, Waterloo, Ontario
  - Innovaderm Research Inc., Montreal, Quebec
  - Centre de Recherche Dermatologique du Quebec metropolitain (CRDQ), Québec, Quebec
  - Centre de Recherche Saint-Louis, Québec, Quebec
  - Diex Research Sherbrooke Inc., Sherbrooke, Quebec
- Germany (6):
  - Fachklinik Bad Bentheim, Fachbereich Dermatologie und Allergologie, Dermatologische Ambulanz, Bad Bentheim
  - Universitaetsklinikum Erlangen Hautklinik Studienambulanz, Erlangen
  - Universitätsklinikum Frankfurt, Klinik für Dermatologie, Venerologie und Allergologie, Frankfurt am Main
  - Universitaetsklinikum Schleswig-Holstein, Campus Luebeck CCIM, Lübeck
  - Universitaetsmedizin der Johannes Gutenberg-Universitaet Mainz, Mainz
  - Universitaetsklinikum Muenster, Münster
- Istituti Fisioterapici Ospitalieri, Istituto di Ricovero e Cura a Carattere Scientifico,, Roma, RM, Italy
- Japan (5):
  - Nagoya City University Hospital - Dermatology, Nagoya, Aichi-ken
  - Tohoku University Hospital, Sendai, Miyagi
  - Nippon Medical School Hospital, Bunkyo-ku, Tokyo
  - Tokyo Medical University Hospital, Shinjuku-ku, Tokyo
  - Yamanashi Prefectural Central Hospital, Kofu, Yamanashi
- South Korea (5):
  - Dongguk University Ilsan Hospital, Goyang-si, Gyeonggi-do
  - The Catholic University of Korea, St. Vincent's Hospital, Suwon, Gyeonggi-do
  - Ajou University Hospital, Suwon, Gyeonggi-do
  - Inha University Hospital, Incheon
  - Severance Hospital, Yonsei University Health System, Seoul
- Spain (5):
  - Hospital de la Santa Creu i Sant Pau, Barcelona
  - Hospital Universitario Reina Sofia, Córdoba
  - Hospital Universitario Ramón y Cajal, Madrid
  - Hospital Universitario La Paz, Madrid
  - Hospital Universitari i Politecnic La Fe, Valencia
- Taiwan (3):
  - Chang Gung Medical Foundation - Kaohsiung Chang Gung Memorial Hospital, Kaohsiung City
  - National Cheng Kung University Hospital, Tainan
  - National Taiwan University Hospital, Taipei

IPD SHARING:
Plan to Share IPD: Yes
Pfizer will provide access to individual de-identified participant data and related study documents (e.g. protocol, Statistical Analysis Plan (SAP), Clinical Study Report (CSR)) upon request from qualified researchers, and subject to certain criteria, conditions, and exceptions. Further details on Pfizer's data sharing criteria and process for requesting access can be found at: https://www.pfizer.com/science/clinical_trials/trial_data_and_results/data_requests.
URL: https://www.pfizer.com/science/clinical_trials/trial_data_and_results/data_requests

REFERENCES:
- [Derived] Yamaguchi Y, Peeva E, Duca ED, Facheris P, Bar J, Shore R, Cox LA, Sloan A, Thaci D, Ganesan A, Han G, Ezzedine K, Ye Z, Guttman-Yassky E. Ritlecitinib, a JAK3/TEC family kinase inhibitor, stabilizes active lesions and repigments stable lesions in vitiligo. Arch Dermatol Res. 2024 Jul 18;316(7):478. doi: 10.1007/s00403-024-03182-y. PMID 39023568
- [Derived] Wojciechowski J, S Purohit V, Huh Y, Banfield C, Nicholas T. Evolution of Ritlecitinib Population Pharmacokinetic Models During Clinical Drug Development. Clin Pharmacokinet. 2023 Dec;62(12):1765-1779. doi: 10.1007/s40262-023-01318-3. Epub 2023 Nov 2. PMID 37917289
- [Derived] Guttman-Yassky E, Del Duca E, Da Rosa JC, Bar J, Ezzedine K, Ye Z, He W, Hyde C, Hassan-Zahraee M, Yamaguchi Y, Peeva E. Improvements in immune/melanocyte biomarkers with JAK3/TEC family kinase inhibitor ritlecitinib in vitiligo. J Allergy Clin Immunol. 2024 Jan;153(1):161-172.e8. doi: 10.1016/j.jaci.2023.09.021. Epub 2023 Sep 28. PMID 37777018
- [Derived] Ezzedine K, Peeva E, Yamaguchi Y, Cox LA, Banerjee A, Han G, Hamzavi I, Ganesan AK, Picardo M, Thaci D, Harris JE, Bae JM, Tsukamoto K, Sinclair R, Pandya AG, Sloan A, Yu D, Gandhi K, Vincent MS, King B. Efficacy and safety of oral ritlecitinib for the treatment of active nonsegmental vitiligo: A randomized phase 2b clinical trial. J Am Acad Dermatol. 2023 Feb;88(2):395-403. doi: 10.1016/j.jaad.2022.11.005. Epub 2022 Nov 9. PMID 36370907
- See also: To obtain contact information for a study center near you, click here. — https://pmiform.com/clinical-trial-info-request?StudyID=B7981019

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: A total of 578 participants were screened for this study; 366 were randomized to treatment and 364 (99.5%) received treatment in the Dose Ranging Period.
Groups:
- PF-06651600 200 mg - 50 mg QD: Participants were randomized to receive ritlecitinib (PF-06651600) induction dose of 200 mg QD for 4 weeks followed by ritlecitinib 50 mg QD for another 20 weeks.
- PF-06651600 100 mg - 50 mg QD: Participants were randomized to receive ritlecitinib induction dose of 100 mg QD for 4 weeks followed by ritlecitinib 50 mg QD for another 20 weeks.
- PF-06651600 50 mg QD: Participants were randomized to receive ritlecitinib 50 mg QD for 24 weeks.
- PF-06651600 30 mg QD: Participants were randomized to receive ritlecitinib 30 mg QD for 24 weeks.
- PF-06651600 10 mg QD: Participants were randomized to receive ritlecitinib 10 mg QD for 24 weeks.
- Placebo: Participants were randomized to receive placebo for 24 weeks.
- Extension (EXT) PF-06700841 60 mg - 30 mg QD: After a 4-week drug holiday, participants received induction dose of brepocitinib (PF-06700841) 60 mg QD for 4 weeks followed by brepocitinib 30 mg QD for 16 weeks. This arm was open label.
- EXT PF-06651600 200 Mg-50 mg QD + nbUVB: Induction dose of ritlecitinib 200 mg QD plus standardized narrow band UVB (nbUVB) add-on therapy for 4 weeks followed by ritlecitinib 50 mg QD plus standardized nbUVB add-on therapy for 20 weeks (only for participants who provided nbUVB consent). Participants who had <10% improvement in percent change in VASI at Extension Week 12 from the baseline value at Dose Ranging Period Week 24 were discontinued from the treatment and entered Follow-up Period. This arm was open label.
- EXT PF-06651600 200 mg - 50 mg QD: Induction dose of ritlecitinib 200 mg QD of for 4 weeks followed by ritlecitinib 50 mg QD for 20 weeks. This arm was double blinded.
- EXT PF-06651600 50 mg QD: Ritlecitinib 50 mg QD for 24 weeks. This arm was double blinded.
- EXT PF-06651600 30 mg QD: Ritlecitinib 30 mg QD of for 24 weeks. This arm was double blinded.
Period: Dose Ranging Period
Arm/Group | PF-06651600 200 mg - 50 mg QD | PF-06651600 100 mg - 50 mg QD | PF-06651600 50 mg QD | PF-06651600 30 mg QD | PF-06651600 10 mg QD | Placebo | Extension (EXT) PF-06700841 60 mg - 30 mg QD | EXT PF-06651600 200 Mg-50 mg QD + nbUVB | EXT PF-06651600 200 mg - 50 mg QD | EXT PF-06651600 50 mg QD | EXT PF-06651600 30 mg QD
Started (The first 6 treatment groups entered this Dose Ranging Period.) | 65 | 67 | 67 | 50 | 49 | 66 | 0 | 0 | 0 | 0 | 0
Completed | 53 | 58 | 54 | 36 | 42 | 55 | 0 | 0 | 0 | 0 | 0
Not Completed | 12 | 9 | 13 | 14 | 7 | 11 | 0 | 0 | 0 | 0 | 0
Not completed — Adverse Event | 2 | 4 | 5 | 2 | 3 | 3 | 0 | 0 | 0 | 0 | 0
Not completed — Lack of Efficacy | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — Lost to Follow-up | 2 | 0 | 1 | 1 | 1 | 2 | 0 | 0 | 0 | 0 | 0
Not completed — Protocol Violation | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — Withdrawal by Subject | 8 | 4 | 3 | 9 | 2 | 3 | 0 | 0 | 0 | 0 | 0
Not completed — Medication Error Without Associated Adverse Event | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — No Longer Meets Eligibility Criteria | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — Other | 0 | 0 | 2 | 0 | 0 | 3 | 0 | 0 | 0 | 0 | 0
Period: Extension Period
Arm/Group | PF-06651600 200 mg - 50 mg QD | PF-06651600 100 mg - 50 mg QD | PF-06651600 50 mg QD | PF-06651600 30 mg QD | PF-06651600 10 mg QD | Placebo | Extension (EXT) PF-06700841 60 mg - 30 mg QD | EXT PF-06651600 200 Mg-50 mg QD + nbUVB | EXT PF-06651600 200 mg - 50 mg QD | EXT PF-06651600 50 mg QD | EXT PF-06651600 30 mg QD
Started (The last 5 EXT treatment groups entered this Extension Period. Three participants were lost to follow-up after completing the Dose Ranging Period, and no extension treatment was recorded for these 3 participants. A total of 295 participants were assigned to the Extension Period, among whom 293 received treatment.) | 0 | 0 | 0 | 0 | 0 | 0 | 55 | 43 | 187 | 6 | 2
Completed | 0 | 0 | 0 | 0 | 0 | 0 | 47 | 27 | 158 | 3 | 2
Not Completed | 0 | 0 | 0 | 0 | 0 | 0 | 8 | 16 | 29 | 3 | 0
Not completed — Adverse Event | 0 | 0 | 0 | 0 | 0 | 0 | 3 | 1 | 6 | 0 | 0
Not completed — Lack of Efficacy | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 9 | 2 | 0 | 0
Not completed — Lost to Follow-up | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0
Not completed — Protocol Violation | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Not completed — Withdrawal by Subject | 0 | 0 | 0 | 0 | 0 | 0 | 3 | 3 | 12 | 3 | 0
Not completed — Medication Error Without Associated Adverse Event | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0
Not completed — No Longer Meets Eligibility Criteria | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Not completed — Other | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 2 | 4 | 0 | 0

BASELINE CHARACTERISTICS:
Population: Baseline analysis population included all participants who received at least 1 dose of randomized study medication and had a baseline and at least 1 post-baseline measurement (after taking randomization study medication).
Groups:
- Total: Total of all reporting groups
Arm/Group | PF-06651600 200 mg - 50 mg QD | PF-06651600 100 mg - 50 mg QD | PF-06651600 50 mg QD | PF-06651600 30 mg QD | PF-06651600 10 mg QD | Placebo | Total
Number analyzed (Participants) | 65 | 67 | 67 | 50 | 49 | 66 | 364
Age, Customized [Count of Participants; unit: Participants]
  <18 Years | 0 | 0 | 0 | 0 | 0 | 0 | 0
  18 - 44 Years | 33 | 29 | 33 | 20 | 16 | 30 | 161
  45 - 64 Years | 30 | 37 | 34 | 30 | 31 | 32 | 194
  ≥65 Years | 2 | 1 | 0 | 0 | 2 | 4 | 9
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 30 | 31 | 39 | 28 | 25 | 40 | 193
  Male | 35 | 36 | 28 | 22 | 24 | 26 | 171
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 11 | 9 | 11 | 12 | 7 | 7 | 57
  Not Hispanic or Latino | 54 | 58 | 54 | 38 | 41 | 58 | 303
  Unknown or Not Reported | 0 | 0 | 2 | 0 | 1 | 1 | 4
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 1 | 0 | 0 | 1
  Asian | 15 | 17 | 17 | 5 | 11 | 21 | 86
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Black or African American | 3 | 0 | 0 | 4 | 1 | 2 | 10
  White | 44 | 47 | 45 | 39 | 33 | 38 | 246
  More than one race | 0 | 1 | 1 | 0 | 2 | 1 | 5
  Unknown or Not Reported | 3 | 2 | 4 | 1 | 2 | 4 | 16

OUTCOME MEASURES:

1. Primary Outcome: Percent Change From Baseline in Central Read Facial-Vitiligo Area Scoring Index (F-VASI) at Week 24 - Dose Ranging (DR) Period
Description: Central read F-VASI was assessed based on the facial photographs taken at the site. Central read F-VASI was calculated using a formula that included contribution of affected facial surface areas showing all 6 different depigmentation rates (0.1, 0.25, 0.5, 0.75, 0.9 and 1) with a modified method: F-VASI (central read)=Ʃ [Affected Facial Surface Area] × 4 × [Depigmentation Rates]. Face was defined as the area from the hairline on top of the forehead to the jawline at the bottom of the cheeks. F-VASI (central read) ranged from 0.000 to 4.000 by defining the affected Facial Surface Area (expressed as the value between 0.0 to 1.0) being 4% of total Body Surface Area. The higher score of F-VASI signified severer symptoms of non-segmental vitiligo. Percent change from baseline in central read F-VASI = ((post-baseline central read F-VASI - baseline central read F-VASI)/baseline central read F-VASI)×100. A negative percent change from baseline in central read F-VASI signified an improvement.
Time Frame: Baseline, Week 24 (Baseline was defined as the last measurement prior to Study Day 18)
Population: The analysis population included all participants who received at least 1 dose of randomized study medication and had a baseline and at least 1 post-baseline measurement (after taking randomization study medication). Number of participants analyzed signifies number of participants who were evaluable for this outcome measure.
Measure: Least Squares Mean (Standard Error); unit: Percent Change
Arm/Group | PF-06651600 200 mg - 50 mg QD | PF-06651600 100 mg - 50 mg QD | PF-06651600 50 mg QD | PF-06651600 30 mg QD | PF-06651600 10 mg QD | Placebo
Number analyzed (Participants) | 62 | 63 | 59 | 45 | 48 | 57
Percent Change | -21.2 (4.13) | -21.2 (4.16) | -18.5 (4.44) | -14.6 (5.47) | -3.0 (4.65) | 2.1 (4.06)
Statistical Analysis 1: Comparison: PF-06651600 200 mg - 50 mg QD vs Placebo; Test type: Superiority; p < 0.0001, ANCOVA — Hochberg's step-up procedure was conducted to compare ritlecitinib 200mg - 50mg QD dose group vs placebo using observed p-values. The familywise Type 1 error rate was controlled at one-sided 0.05. Hochberg adjusted p-value is presented here; Least Squares Mean Difference (Net) = -23.2, 90% CI 2-sided [-32.53 to -13.96], Standard Error of Mean 5.62
Statistical Analysis 2: Comparison: PF-06651600 100 mg - 50 mg QD vs Placebo; Test type: Superiority; p < 0.0001, ANCOVA — Hochberg's step-up procedure was conducted to compare ritlecitinib 100mg - 50mg QD dose group vs placebo using observed p-values. The familywise Type 1 error rate was controlled at one-sided 0.05. Hochberg adjusted p-value is presented here; Least Squares Mean Difference (Net) = -23.2, 90% CI 2-sided [-32.53 to -13.93], Standard Error of Mean 5.63
Statistical Analysis 3: Comparison: PF-06651600 50 mg QD vs Placebo; Test type: Superiority; p = 0.0003, ANCOVA — Hochberg's step-up procedure was conducted to compare the ritlecitinib 50 mg QD dose group vs placebo using observed p-values. The familywise Type 1 error rate was controlled at one-sided 0.05. Hochberg adjusted p-value is presented here; Least Squares Mean Difference (Net) = -20.6, 90% CI 2-sided [-30.23 to -10.93], Standard Error of Mean 5.84
Statistical Analysis 4: Comparison: PF-06651600 30 mg QD vs Placebo; Test type: Superiority; p = 0.0068, ANCOVA — Hochberg's step-up procedure was conducted to compare the ritlecitinib 30 mg QD dose group vs placebo using observed p-values. The familywise Type 1 error rate was controlled at one-sided 0.05. One-sided unadjusted p-value is presented here; Least Squares Mean Difference (Net) = -16.7, 90% CI 2-sided [-27.77 to -5.61], Standard Error of Mean 6.71
Statistical Analysis 5: Comparison: PF-06651600 10 mg QD; Test type: Superiority; p = 0.2015, ANCOVA — Hochberg's step-up procedure was conducted to compare the ritlecitinib 10 mg QD dose group vs placebo using observed p-values. The familywise Type 1 error rate was controlled at one-sided 0.05. One-sided unadjusted p-value is presented here; Least Squares Mean Difference (Net) = -5.1, 90% CI 2-sided [-15.02 to 4.91], Standard Error of Mean 6.03

2. Secondary Outcome: Percentage of Participants Achieving Central F-VASI75 at Week 24 - DR Period
Description: This outcome measure was the percentage of participants achieving at least 75% improvement from baseline in central read F-VASI (F-VASI75) at Week 24. A negative percent change from baseline in central read F-VASI signified an improvement. The central read F-VASI75 response rate was analyzed by first treating the missing data (non-COVID-19 related) as non responders and then applying Chan and Zhang exact confidence interval (CI) method at Week 24.
  Central read F-VASI75=1 if percent change from baseline ≥75; central read F-VASI75=0 if percent change from baseline <75. Percent change from baseline in F-VASI=((post-baseline F-VASI - baseline F-VASI)/baseline F-VASI)×100. Baseline was defined as the last measurement prior to study Day 18.
Time Frame: Week 24
Population: as for outcome 1
Measure: Number; unit: Percentage of Participants
Arm/Group | PF-06651600 200 mg - 50 mg QD | PF-06651600 100 mg - 50 mg QD | PF-06651600 50 mg QD | PF-06651600 30 mg QD | PF-06651600 10 mg QD | Placebo
Number analyzed (Participants) | 58 | 59 | 52 | 37 | 43 | 57
Percentage of Participants | 12.1 | 8.5 | 7.7 | 2.7 | 2.3 | 0

3. Secondary Outcome: Percentage of Participants Achieving T-VASI50 at Week 24 - DR Period
Description: Total body VASI (T-VASI) was calculated using a formula that included contribution from 6 different body regions (possible range, 0-100) with a modified method: T-VASI= Ʃ[Hand Units]×[Depigmentation]. One hand unit, which encompassed the palm plus the volar surface of all the digits, was approximately 1% of the total body surface area and was used as a guide to estimate the baseline percentage of vitiligo involvement of each body region. The body was divided into 6 separate and mutually exclusive regions: face/neck, hands, upper extremities (excluding hands), trunk, lower extremities (excluding feet), and feet. The extent of depigmentation was expressed by percentages: 0, 10%, 25%, 50%, 75%, 90% or 100%. The data below was the percentage of participants achieving at least 50% improvement from baseline in T-VASI (T-VASI50) at Week 24. Negative percent change from baseline in T-VASI signified an improvement. Baseline was defined as the last measurement prior to first dosing (Day 1).
Time Frame: Week 24
Population: as for outcome 1
Measure: Number; unit: Percentage of Participants
Groups:
- PF-06651600 200mg - 50mg QD: Participants were randomized to receive ritlecitinib induction dose (200 mg QD) for 4 weeks followed by maintenance dosing of 50 mg QD for 20 weeks
Arm/Group | PF-06651600 200mg - 50mg QD | PF-06651600 100 mg - 50 mg QD | PF-06651600 50 mg QD | PF-06651600 30 mg QD | PF-06651600 10 mg QD | Placebo
Number analyzed (Participants) | 63 | 65 | 65 | 47 | 49 | 66
Percentage of Participants | 7.9 | 4.6 | 4.6 | 10.6 | 4.1 | 9.1

4. Secondary Outcome: Percent Change From Baseline in T-VASI at Designated Time Points - DR Period
Description: The T-VASI was calculated using a formula that included contribution from 6 different body regions (possible range, 0-100) with a modified method: VASI = Ʃ [Hand Units] × [Depigmentation]. One hand unit, which encompassed the palm plus the volar surface of all the digits, was approximately 1% of the total body surface area and was used as a guide to estimate the baseline percentage of vitiligo involvement of each body region. The body was divided into 6 separate and mutually exclusive regions: face/neck, hands, upper extremities (excluding hands), trunk, lower extremities (excluding the feet), and feet. The extent of depigmentation was expressed by the following percentages: 0, 10%, 25%, 50%, 75%, 90%, or 100%. Percent change from baseline in T-VASI=((post-baseline T-VASI - baseline T-VASI)/baseline T-VASI)×100. Negative percent change from baseline in T-VASI signified an improvement. Baseline was defined as the last measurement prior to first dosing (Day 1).
Time Frame: Baseline, Weeks 4, 8, 12, 16, 20 and 24
Population: The analysis population included all participants who received at least 1 dose of randomized study medication and had a baseline and at least 1 post-baseline measurement (after taking randomization study medication). Number of participants analyzed signifies number of participants who were evaluable for this outcome measure. Number analyzed refers to number of participants evaluable for specified rows of categories.
Measure: Least Squares Mean (Standard Error); unit: Percent Change
Arm/Group | PF-06651600 200mg - 50mg QD | PF-06651600 100 mg - 50 mg QD | PF-06651600 50 mg QD | PF-06651600 30 mg QD | PF-06651600 10 mg QD | Placebo
Number analyzed (Participants) | 64 | 67 | 67 | 50 | 49 | 66
Percent Change
  Week 4: number analyzed (Participants) | 64 | 66 | 64 | 50 | 47 | 63
  Week 4 | -2.4 (1.51) | -3.0 (1.50) | -2.6 (1.50) | -5.1 (1.72) | -2.9 (1.76) | -1.4 (1.52)
  Week 8: number analyzed (Participants) | 63 | 65 | 63 | 48 | 48 | 64
  Week 8 | -6.2 (2.03) | -5.4 (2.01) | -5.1 (2.01) | -6.6 (2.33) | -3.0 (2.32) | -5.8 (2.02)
  Week 12: number analyzed (Participants) | 59 | 62 | 60 | 44 | 46 | 61
  Week 12 | -7.2 (2.44) | -11.9 (2.40) | -9.1 (2.40) | -11.4 (2.82) | -4.9 (2.76) | -8.0 (2.40)
  Week 16: number analyzed (Participants) | 56 | 57 | 55 | 43 | 43 | 58
  Week 16 | -10.0 (2.66) | -13.1 (2.67) | -12.6 (2.66) | -11.9 (3.03) | -5.7 (3.03) | -12.0 (2.62)
  Week 20: number analyzed (Participants) | 52 | 59 | 53 | 43 | 41 | 55
  Week 20 | -13.8 (3.13) | -16.0 (2.98) | -14.2 (3.07) | -12.0 (3.43) | -9.2 (3.51) | -13.3 (3.04)
  Week 24: number analyzed (Participants) | 52 | 58 | 52 | 36 | 41 | 56
  Week 24 | -14.7 (3.49) | -19.2 (3.29) | -14.7 (3.44) | -14.0 (4.15) | -12.1 (3.88) | -11.0 (3.34)

5. Secondary Outcome: Percent Change From Baseline in Central Read F-VASI at Designated Time Points - DR Period
Description: The central read F-VASI was assessed based on the facial photographs taken at the site. The central read F-VASI was calculated using a formula that included contribution of affected facial surface areas showing all 6 different depigmentation rates (0.1, 0.25, 0.5, 0.75, 0.9 and 1) with a modified method: F-VASI (central read)=Ʃ [Affected Facial Surface Area] × 4 × [Depigmentation Rates]. Face was defined as the area from the hairline on top of the forehead to the jawline at the bottom of the cheeks. F-VASI (central read) ranged from 0.000 to 4.000 by defining the affected Facial Surface Area (expressed as the value between 0.0 to 1.0) being 4% of total Body Surface Area.
  Percent change from baseline in central read F-VASI = ((post-baseline central read F-VASI - baseline central read F-VASI)/baseline central read F-VASI)×100. Negative percent change from baseline in F-VASI signified an improvement. Baseline was defined as the last measurement prior to Study Day 18.
Time Frame: Baseline, Weeks 4, 8, 16 and 24
Population: as for outcome 4
Measure: Least Squares Mean (Standard Error); unit: Percent Change
Arm/Group | PF-06651600 200mg - 50mg QD | PF-06651600 100 mg - 50 mg QD | PF-06651600 50 mg QD | PF-06651600 30 mg QD | PF-06651600 10 mg QD | Placebo
Number analyzed (Participants) | 62 | 63 | 59 | 45 | 48 | 57
Percent Change
  Week 4: number analyzed (Participants) | 61 | 60 | 55 | 44 | 47 | 56
  Week 4 | 0.1 (0.80) | 0.4 (0.82) | -0.2 (0.84) | -1.2 (0.94) | 0.0 (0.91) | 0.6 (0.83)
  Week 8: number analyzed (Participants) | 57 | 57 | 52 | 43 | 47 | 55
  Week 8 | -7.0 (1.42) | -5.3 (1.44) | -1.8 (1.46) | -1.4 (1.62) | -0.1 (1.55) | -0.2 (1.44)
  Week 16: number analyzed (Participants) | 51 | 49 | 49 | 34 | 37 | 47
  Week 16 | -17.0 (3.16) | -16.4 (3.25) | -10.7 (3.19) | -13.3 (3.87) | -5.6 (3.67) | -0.2 (3.27)
  Week 24: number analyzed (Participants) | 49 | 49 | 41 | 27 | 37 | 50
  Week 24 | -21.2 (4.13) | -21.2 (4.16) | -18.5 (4.44) | -14.6 (5.47) | -3.0 (4.65) | 2.1 (4.06)

6. Secondary Outcome: Percent Change From Baseline in Local F-VASI at Designated Time Points - DR Period
Description: The site assessment of the F-VASI was calculated using a formula that included contribution from face (possible range, 0.00 4.00): Local F-VASI = [Digit Units] × [Depigmentation] × 0.1. Scalp, neck, eyebrows, eyelashes, and vermilion were excluded from this calculation. The volar surface of 1 digit (the participant's thumb) was approximately 0.1% of the total body surface area and was used as a guide to estimate the baseline percentage of vitiligo involvement of face. The extent of depigmentation was expressed by the following percentages: 0, 10%, 25%, 50%, 75%, 90%, or 100%.
  Percent change from baseline in Local F-VASI = ((post baseline Local F-VASI - baseline Local F-VASI)/baseline Local F-VASI)×100. Negative percent change from baseline in F-VASI signified an improvement. Baseline was defined as the last measurement prior to first dosing (Day 1).
Time Frame: Baseline, Weeks 4, 8, 12, 16, 20 and 24
Population: as for outcome 4
Measure: Least Squares Mean (Standard Error); unit: Percent Change
Arm/Group | PF-06651600 200mg - 50mg QD | PF-06651600 100 mg - 50 mg QD | PF-06651600 50 mg QD | PF-06651600 30 mg QD | PF-06651600 10 mg QD | Placebo
Number analyzed (Participants) | 64 | 67 | 67 | 50 | 49 | 66
Percent Change
  Week 4: number analyzed (Participants) | 64 | 66 | 64 | 50 | 47 | 63
  Week 4 | -4.9 (2.63) | 3.1 (2.61) | -5.0 (2.60) | 0.4 (2.96) | -5.3 (3.05) | -6.3 (2.63)
  Week 8: number analyzed (Participants) | 63 | 65 | 63 | 48 | 48 | 64
  Week 8 | -11.3 (5.35) | 0.4 (5.32) | -8.8 (5.30) | 10.1 (6.09) | -7.3 (6.12) | -7.5 (5.31)
  Week 12: number analyzed (Participants) | 59 | 62 | 60 | 44 | 46 | 61
  Week 12 | -15.9 (4.16) | -6.5 (4.11) | -12.2 (4.10) | -7.1 (4.77) | -9.8 (4.72) | -11.4 (4.08)
  Week 16: number analyzed (Participants) | 56 | 57 | 56 | 43 | 44 | 58
  Week 16 | -19.4 (4.85) | -6.2 (4.88) | -19.7 (4.82) | -6.4 (5.48) | -10.3 (5.46) | -13.3 (4.75)
  Week 20: number analyzed (Participants) | 52 | 59 | 53 | 43 | 41 | 55
  Week 20 | -21.9 (5.59) | -12.9 (5.35) | -23.2 (5.52) | 0.0 (6.11) | -14.4 (6.30) | -15.3 (5.44)
  Week 24: number analyzed (Participants) | 52 | 58 | 52 | 36 | 41 | 56
  Week 24 | -28.3 (5.70) | -20.6 (5.38) | -26.2 (5.61) | -4.3 (6.70) | -13.9 (6.32) | -18.1 (5.43)

7. Secondary Outcome: Percent Change From Baseline in SA-VES at Designated Time Points - DR Period
Description: The Self-Assessment Vitiligo Extent Score (SA-VES) was a validated patient report outcome measurement instrument to provide information about disease extent. Vitiligo Extent Score (VES) was a measure to express the overall vitiligo involvement of the body (extent). Clinical illustrations for 19 separate body areas that reflected different degrees of involvement (1%, 5%, 10%, 25%, 50% and 75% depigmentation) were chosen to represent the participant's skin lesions to get the total extent of the disease. VES was a sum of all surface measurement that was similar to VASI. Baseline was defined as the last measurement prior to first dosing (Day 1).
Time Frame: Baseline, Weeks 4, 16 and 24
Population: as for outcome 4
Measure: Least Squares Mean (Standard Error); unit: Percent Change
Arm/Group | PF-06651600 200mg - 50mg QD | PF-06651600 100 mg - 50 mg QD | PF-06651600 50 mg QD | PF-06651600 30 mg QD | PF-06651600 10 mg QD | Placebo
Number analyzed (Participants) | 64 | 67 | 67 | 50 | 49 | 66
Percent Change
  Week 4: number analyzed (Participants) | 62 | 66 | 64 | 50 | 47 | 63
  Week 4 | 2.7 (17.19) | 1.1 (16.71) | -1.1 (16.74) | 4.9 (19.25) | 4.9 (19.84) | 50.4 (17.13)
  Week 16: number analyzed (Participants) | 54 | 55 | 56 | 41 | 44 | 58
  Week 16 | 4.7 (13.82) | -0.5 (13.48) | -3.7 (13.45) | 6.9 (15.53) | -0.5 (15.87) | 52.5 (13.72)
  Week 24: number analyzed (Participants) | 50 | 56 | 49 | 32 | 40 | 55
  Week 24 | 0.0 (10.35) | -3.5 (10.02) | -4.3 (10.11) | -4.4 (11.89) | -1.6 (11.77) | 44.0 (10.16)

8. Secondary Outcome: Absolute Change From Baseline in T-VASI at Designated Time Points - DR Period
Description: The T-VASI was calculated using a formula that included contribution from 6 different body regions (possible range, 0-100) with a modified method: VASI = Ʃ [Hand Units] × [Depigmentation]. One hand unit, which encompassed the palm plus the volar surface of all the digits, was approximately 1% of the total body surface area and was used as a guide to estimate the baseline percentage of vitiligo involvement of each body region. The body was divided into 6 separate and mutually exclusive regions: face/neck, hands, upper extremities (excluding hands), trunk, lower extremities (excluding the feet), and feet. The extent of depigmentation was expressed by the following percentages: 0, 10%, 25%, 50%, 75%, 90%, or 100%.
  The absolute change from baseline in T-VASI was analyzed using the ANCOVA analysis. Negative change from baseline in T-VASI signified an improvement. Baseline was defined as the last measurement prior to first dosing (Day 1).
Time Frame: Baseline, Weeks 4, 8, 12, 16, 20 and 24
Population: The analysis population included all participants who received at least 1 dose of randomized study medication and have a baseline and at least 1 post-baseline measurement (after taking randomization study medication). Number of participants analyzed signifies number of participants who were evaluable for this outcome measure. Number analyzed refers to number of participants evaluable for specified rows of categories.
Measure: Least Squares Mean (Standard Error); unit: Units on a Scale
Arm/Group | PF-06651600 200mg - 50mg QD | PF-06651600 100 mg - 50 mg QD | PF-06651600 50 mg QD | PF-06651600 30 mg QD | PF-06651600 10 mg QD | Placebo
Number analyzed (Participants) | 64 | 67 | 67 | 50 | 49 | 66
Units on a Scale
  Week 4: number analyzed (Participants) | 64 | 66 | 64 | 50 | 47 | 63
  Week 4 | -0.3 (0.25) | -0.5 (0.25) | -0.6 (0.25) | -1.0 (0.28) | -0.4 (0.29) | -0.2 (0.25)
  Week 8: number analyzed (Participants) | 63 | 65 | 63 | 48 | 48 | 64
  Week 8 | -0.9 (0.32) | -0.9 (0.32) | -0.9 (0.32) | -1.2 (0.37) | -0.5 (0.36) | -0.9 (0.32)
  Week 12: number analyzed (Participants) | 59 | 62 | 60 | 44 | 46 | 61
  Week 12 | -1.1 (0.41) | -2.0 (0.40) | -1.6 (0.40) | -1.8 (0.47) | -0.9 (0.46) | -1.6 (0.40)
  Week 16: number analyzed (Participants) | 56 | 57 | 55 | 43 | 43 | 58
  Week 16 | -1.5 (0.46) | -2.1 (0.46) | -1.9 (0.46) | -1.9 (0.53) | -0.9 (0.53) | -2.2 (0.46)
  Week 20: number analyzed (Participants) | 52 | 59 | 53 | 43 | 41 | 55
  Week 20 | -2.0 (0.55) | -2.8 (0.53) | -2.3 (0.54) | -2.0 (0.61) | -1.7 (0.62) | -2.2 (0.54)
  Week 24: number analyzed (Participants) | 52 | 58 | 52 | 36 | 41 | 56
  Week 24 | -2.3 (0.62) | -3.4 (0.59) | -2.4 (0.61) | -2.7 (0.74) | -2.0 (0.69) | -1.8 (0.60)

9. Secondary Outcome: Percentage of Participants Achieving T-VASI50 at Designated Time Points - DR Period
Description: T-VASI was calculated by a formula that included contribution from 6 body regions (possible range, 0-100): T-VASI = Ʃ [Hand Units] × [Depigmentation]. One hand unit, which encompassed the palm plus the volar surface of all the digits, was approximately 1% of the total body surface area and was used as a guide to estimate the baseline percentage of vitiligo involvement of each body region. The body was divided into 6 mutually exclusive regions: face/neck, hands, upper extremities, trunk, lower extremities, and feet. The extent of depigmentation was expressed by the percentages: 0, 10%, 25%, 50%, 75%, 90% or 100%. The outcome measure was the percentage of participants achieving at least 50% improvement from baseline in T-VASI (T-VASI50). Percent change from baseline in T-VASI=((post-baseline T-VASI - baseline T-VASI)/baseline T-VASI)×100. Negative percent change from baseline in T-VASI signified an improvement. Baseline was defined as the last measurement prior to first dosing (Day 1).
Time Frame: Baseline, Weeks 4, 8, 12, 16, 20 and 24
Population: as for outcome 4
Measure: Number; unit: Percentage of Participants
Arm/Group | PF-06651600 200mg - 50mg QD | PF-06651600 100 mg - 50 mg QD | PF-06651600 50 mg QD | PF-06651600 30 mg QD | PF-06651600 10 mg QD | Placebo
Number analyzed (Participants) | 64 | 67 | 67 | 50 | 49 | 66
Percentage of Participants
  Week 4 | 1.6 | 1.5 | 0 | 2.0 | 0 | 0
  Week 8 | 1.6 | 1.5 | 1.5 | 4.0 | 0 | 1.5
  Week 12: number analyzed (Participants) | 62 | 66 | 66 | 49 | 48 | 66
  Week 12 | 1.6 | 1.5 | 1.5 | 4.1 | 0 | 4.5
  Week 16: number analyzed (Participants) | 63 | 62 | 66 | 47 | 46 | 63
  Week 16 | 0 | 3.2 | 0 | 2.1 | 0 | 6.3
  Week 20: number analyzed (Participants) | 61 | 67 | 64 | 49 | 48 | 63
  Week 20 | 4.9 | 1.5 | 1.6 | 6.1 | 2.1 | 9.5
  Week 24: number analyzed (Participants) | 63 | 65 | 65 | 47 | 49 | 66
  Week 24 | 7.9 | 4.6 | 4.6 | 10.6 | 4.1 | 9.1

10. Secondary Outcome: Percentage of Participants Achieving T-VASI75 at Designated Time Points - DR Period
Description: T-VASI was calculated by a formula that included contribution from 6 body regions (possible range, 0-100): T-VASI = Ʃ [Hand Units] × [Depigmentation]. One hand unit, which encompassed the palm plus the volar surface of all the digits, was approximately 1% of the total body surface area and was used as a guide to estimate the baseline percentage of vitiligo involvement of each body region. The body was divided into 6 mutually exclusive regions: face/neck, hands, upper extremities, trunk, lower extremities, and feet. The extent of depigmentation was expressed by the percentages: 0, 10%, 25%, 50%, 75%, 90% or 100%. The outcome measure was the percentage of participants achieving at least 75% improvement from baseline in T-VASI (T-VASI75). Percent change from baseline in T-VASI=((post-baseline T-VASI - baseline T-VASI)/baseline T-VASI)×100. Negative percent change from baseline in T-VASI signified an improvement. Baseline was defined as the last measurement prior to first dosing (Day 1).
Time Frame: Baseline, Weeks 4, 8, 12, 16, 20 and 24
Population: as for outcome 4
Measure: Number; unit: Percentage of Participants
Arm/Group | PF-06651600 200mg - 50mg QD | PF-06651600 100 mg - 50 mg QD | PF-06651600 50 mg QD | PF-06651600 30 mg QD | PF-06651600 10 mg QD | Placebo
Number analyzed (Participants) | 64 | 67 | 67 | 50 | 49 | 66
Percentage of Participants
  Week 4 | 0 | 0 | 0 | 0 | 0 | 0
  Week 8 | 0 | 0 | 0 | 0 | 0 | 0
  Week 12: number analyzed (Participants) | 62 | 66 | 66 | 49 | 48 | 66
  Week 12 | 0 | 0 | 0 | 0 | 0 | 0
  Week 16: number analyzed (Participants) | 63 | 62 | 66 | 47 | 46 | 63
  Week 16 | 0 | 0 | 0 | 0 | 0 | 0
  Week 20: number analyzed (Participants) | 61 | 67 | 64 | 49 | 48 | 63
  Week 20 | 0 | 0 | 0 | 0 | 0 | 0
  Week 24: number analyzed (Participants) | 63 | 65 | 65 | 47 | 49 | 66
  Week 24 | 0 | 0 | 0 | 0 | 0 | 0

11. Secondary Outcome: Percentage of Participants Achieving T-VASI90 at Designated Time Points - DR Period
Description: T-VASI was calculated by a formula that included contribution from 6 body regions (possible range, 0-100): T-VASI = Ʃ [Hand Units] × [Depigmentation]. One hand unit, which encompassed the palm plus the volar surface of all the digits, was approximately 1% of the total body surface area and was used as a guide to estimate the baseline percentage of vitiligo involvement of each body region. The body was divided into 6 mutually exclusive regions: face/neck, hands, upper extremities, trunk, lower extremities, and feet. The extent of depigmentation was expressed by the percentages: 0, 10%, 25%, 50%, 75%, 90% or 100%. The outcome measure was the percentage of participants achieving at least 90% improvement from baseline in T-VASI (T-VASI90). Percent change from baseline in T-VASI=((post-baseline T-VASI - baseline T-VASI)/baseline T-VASI)×100. Negative percent change from baseline in T-VASI signified an improvement. Baseline was defined as the last measurement prior to first dosing (Day 1).
Time Frame: Baseline, Weeks 4, 8, 12, 16, 20 and 24
Population: as for outcome 4
Measure: Number; unit: Percentage of Participants
Arm/Group | PF-06651600 200mg - 50mg QD | PF-06651600 100 mg - 50 mg QD | PF-06651600 50 mg QD | PF-06651600 30 mg QD | PF-06651600 10 mg QD | Placebo
Number analyzed (Participants) | 64 | 67 | 67 | 50 | 49 | 66
Percentage of Participants
  Week 4 | 0 | 0 | 0 | 0 | 0 | 0
  Week 8 | 0 | 0 | 0 | 0 | 0 | 0
  Week 12: number analyzed (Participants) | 62 | 66 | 66 | 49 | 48 | 66
  Week 12 | 0 | 0 | 0 | 0 | 0 | 0
  Week 16: number analyzed (Participants) | 63 | 62 | 66 | 47 | 46 | 63
  Week 16 | 0 | 0 | 0 | 0 | 0 | 0
  Week 20: number analyzed (Participants) | 61 | 67 | 64 | 49 | 48 | 63
  Week 20 | 0 | 0 | 0 | 0 | 0 | 0
  Week 24: number analyzed (Participants) | 63 | 65 | 65 | 47 | 49 | 66
  Week 24 | 0 | 0 | 0 | 0 | 0 | 0

12. Secondary Outcome: Percentage of Participants Achieving T-VASI100 at Designated Time Points - DR Period
Description: T-VASI was calculated using a formula that included contribution from 6 body regions (possible range, 0-100): T-VASI = Ʃ [Hand Units] × [Depigmentation]. One hand unit, which encompassed the palm plus the volar surface of all the digits, was approximately 1% of the total body surface area and was used as a guide to estimate the baseline percentage of vitiligo involvement of each body region. The body was divided into 6 mutually exclusive regions: face/neck, hands, upper extremities, trunk, lower extremities, and feet. The extent of depigmentation was expressed by the percentages: 0, 10%, 25%, 50%, 75%, 90% or 100%. This outcome measure was the percentage of participants achieving 100% improvement from baseline in T-VASI (T-VASI100). Percent change from baseline in T-VASI = ((post-baseline T-VASI - baseline T-VASI)/baseline T-VASI)×100. Negative percent change from baseline in T-VASI signified an improvement. Baseline was defined as the last measurement prior to first dosing (Day 1).
Time Frame: Baseline, Weeks 4, 8, 12, 16, 20 and 24
Population: as for outcome 4
Measure: Number; unit: Percentage of Participants
Arm/Group | PF-06651600 200mg - 50mg QD | PF-06651600 100 mg - 50 mg QD | PF-06651600 50 mg QD | PF-06651600 30 mg QD | PF-06651600 10 mg QD | Placebo
Number analyzed (Participants) | 64 | 67 | 67 | 50 | 49 | 66
Percentage of Participants
  Week 4 | 0 | 0 | 0 | 0 | 0 | 0
  Week 8 | 0 | 0 | 0 | 0 | 0 | 0
  Week 12: number analyzed (Participants) | 62 | 66 | 66 | 49 | 48 | 66
  Week 12 | 0 | 0 | 0 | 0 | 0 | 0
  Week 16: number analyzed (Participants) | 63 | 62 | 66 | 47 | 46 | 63
  Week 16 | 0 | 0 | 0 | 0 | 0 | 0
  Week 20: number analyzed (Participants) | 61 | 67 | 64 | 49 | 48 | 63
  Week 20 | 0 | 0 | 0 | 0 | 0 | 0
  Week 24: number analyzed (Participants) | 63 | 65 | 65 | 47 | 49 | 66
  Week 24 | 0 | 0 | 0 | 0 | 0 | 0

13. Secondary Outcome: Percentage of Participants Achieving Central Read F-VASI50 at Designated Time Points - DR Period
Description: The central read F-VASI was calculated using a formula that included contribution of affected facial surface areas showing all 6 different depigmentation rates (0.1, 0.25, 0.5, 0.75, 0.9 and 1) with a modified method: F-VASI (central read)=Ʃ [Affected Facial Surface Area] × 4 × [Depigmentation Rates]. Face was defined as the area from the hairline on top of the forehead to the jawline at the bottom of the cheeks. F-VASI (central read) ranged from 0.000 to 4.000 by defining the affected Facial Surface Area (expressed as the value between 0.0 to 1.0) being 4% of total Body Surface Area. Percent change from baseline in F-VASI = ((post-baseline F-VASI - baseline F-VASI)/baseline F-VASI)×100. This outcome measure was the percentage of participants achieving at least 50% improvement in central read F-VASI from baseline (F-VASI50). Negative percent change from baseline in F-VASI signified an improvement. Baseline was defined as the last measurement prior to Study Day 18.
Time Frame: Baseline, Weeks 4, 8, 16 and 24
Population: as for outcome 4
Measure: Number; unit: Percentage of Participants
Arm/Group | PF-06651600 200mg - 50mg QD | PF-06651600 100 mg - 50 mg QD | PF-06651600 50 mg QD | PF-06651600 30 mg QD | PF-06651600 10 mg QD | Placebo
Number analyzed (Participants) | 62 | 63 | 59 | 45 | 48 | 57
Percentage of Participants
  Week 4 | 0 | 0 | 0 | 2.2 | 0 | 0
  Week 8 | 3.2 | 0 | 0 | 2.2 | 0 | 0
  Week 16: number analyzed (Participants) | 61 | 58 | 58 | 39 | 42 | 52
  Week 16 | 14.8 | 13.8 | 6.9 | 10.3 | 2.4 | 1.9
  Week 24: number analyzed (Participants) | 58 | 59 | 52 | 37 | 43 | 57
  Week 24 | 22.4 | 25.4 | 15.4 | 18.9 | 7.0 | 1.8

14. Secondary Outcome: Percentage of Participants Achieving Central Read F-VASI75 at Designated Time Points - DR Period
Description: The central read F-VASI was calculated using a formula that included contribution of affected facial surface areas showing all 6 different depigmentation rates (0.1, 0.25, 0.5, 0.75, 0.9 and 1) with a modified method: F-VASI (central read)=Ʃ [Affected Facial Surface Area] × 4 × [Depigmentation Rates]. Face was defined as the area from the hairline on top of the forehead to the jawline at the bottom of the cheeks. F-VASI (central read) ranged from 0.000 to 4.000 by defining the affected Facial Surface Area (expressed as the value between 0.0 to 1.0) being 4% of total Body Surface Area. Percent change from baseline in F-VASI = ((post-baseline F-VASI - baseline F-VASI)/baseline F-VASI)×100. This outcome measure was the percentage of participants achieving at least 75% improvement in central read F-VASI from baseline (F-VASI75). Negative percent change from baseline in F-VASI signified an improvement. Baseline was defined as the last measurement prior to Study Day 18.
Time Frame: Baseline, Weeks 4, 8, 16 and 24
Population: as for outcome 4
Measure: Number; unit: Percentage of Participants
Arm/Group | PF-06651600 200mg - 50mg QD | PF-06651600 100 mg - 50 mg QD | PF-06651600 50 mg QD | PF-06651600 30 mg QD | PF-06651600 10 mg QD | Placebo
Number analyzed (Participants) | 62 | 63 | 59 | 45 | 48 | 57
Percentage of Participants
  Week 4 | 0 | 0 | 0 | 0 | 0 | 0
  Week 8 | 0 | 0 | 0 | 0 | 0 | 0
  Week 16: number analyzed (Participants) | 61 | 58 | 58 | 39 | 42 | 52
  Week 16 | 1.6 | 1.7 | 5.2 | 2.6 | 2.4 | 0
  Week 24: number analyzed (Participants) | 58 | 59 | 52 | 37 | 43 | 57
  Week 24 | 12.1 | 8.5 | 7.7 | 2.7 | 2.3 | 0

15. Secondary Outcome: Percentage of Participants Achieving Central Read F-VASI90 at Designated Time Points - DR Period
Description: The central read F-VASI was calculated using a formula that included contribution of affected facial surface areas showing all 6 different depigmentation rates (0.1, 0.25, 0.5, 0.75, 0.9 and 1) with a modified method: F-VASI (central read)=Ʃ [Affected Facial Surface Area] × 4 × [Depigmentation Rates]. Face was defined as the area from the hairline on top of the forehead to the jawline at the bottom of the cheeks. F-VASI (central read) ranged from 0.000 to 4.000 by defining the affected Facial Surface Area (expressed as the value between 0.0 to 1.0) being 4% of total Body Surface Area. Percent change from baseline in F-VASI = ((post-baseline F-VASI - baseline F-VASI)/baseline F-VASI)×100. This outcome measure was the percentage of participants achieving at least 90% improvement in central read F-VASI from baseline (F-VASI90). Negative percent change from baseline in F-VASI signified an improvement. Baseline was defined as the last measurement prior to Study Day 18.
Time Frame: Baseline, Weeks 4, 8, 16 and 24
Population: as for outcome 4
Measure: Number; unit: Percentage of Participants
Arm/Group | PF-06651600 200mg - 50mg QD | PF-06651600 100 mg - 50 mg QD | PF-06651600 50 mg QD | PF-06651600 30 mg QD | PF-06651600 10 mg QD | Placebo
Number analyzed (Participants) | 62 | 63 | 59 | 45 | 48 | 57
Percentage of Participants
  Week 4 | 0 | 0 | 0 | 0 | 0 | 0
  Week 8 | 0 | 0 | 0 | 0 | 0 | 0
  Week 16: number analyzed (Participants) | 61 | 58 | 58 | 39 | 42 | 52
  Week 16 | 0 | 0 | 1.7 | 0 | 0 | 0
  Week 24: number analyzed (Participants) | 58 | 59 | 52 | 37 | 43 | 57
  Week 24 | 1.7 | 0 | 3.8 | 0 | 0 | 0

16. Secondary Outcome: Percentage of Participants Achieving Central Read F-VASI100 at Designated Time Points - DR Period
Description: The central read F-VASI was calculated using a formula that included contribution of affected facial surface areas showing all 6 different depigmentation rates (0.1, 0.25, 0.5, 0.75, 0.9 and 1) with a modified method: F-VASI (central read)=Ʃ [Affected Facial Surface Area] × 4 × [Depigmentation Rates]. Face was defined as the area from the hairline on top of the forehead to the jawline at the bottom of the cheeks. F-VASI (central read) ranged from 0.000 to 4.000 by defining the affected Facial Surface Area (expressed as the value between 0.0 to 1.0) being 4% of total Body Surface Area. Percent change from baseline in F-VASI = ((post-baseline F-VASI - baseline F-VASI)/baseline F-VASI)×100. This outcome measure was the percentage of participants achieving at least 100% improvement in central read F-VASI from baseline (F-VASI100). Negative percent change from baseline in F-VASI signified an improvement. Baseline was defined as the last measurement prior to Study Day 18.
Time Frame: Baseline, Weeks 4, 8, 16 and 24
Population: as for outcome 4
Measure: Number; unit: Percentage of Participants
Arm/Group | PF-06651600 200mg - 50mg QD | PF-06651600 100 mg - 50 mg QD | PF-06651600 50 mg QD | PF-06651600 30 mg QD | PF-06651600 10 mg QD | Placebo
Number analyzed (Participants) | 62 | 63 | 59 | 45 | 48 | 57
Percentage of Participants
  Week 4 | 0 | 0 | 0 | 0 | 0 | 0
  Week 8 | 0 | 0 | 0 | 0 | 0 | 0
  Week 16: number analyzed (Participants) | 61 | 58 | 58 | 39 | 42 | 52
  Week 16 | 0 | 0 | 0 | 0 | 0 | 0
  Week 24: number analyzed (Participants) | 58 | 59 | 52 | 37 | 43 | 57
  Week 24 | 0 | 0 | 0 | 0 | 0 | 0

17. Secondary Outcome: Percentage of Participants Achieving Local F-VASI50 at Designated Time Points - DR Period
Description: The site assessment of the F-VASI was calculated using a formula that included contribution from face (possible range, 0-4): Local F-VASI = [Digit Units] × [Depigmentation] × 0.1. Scalp, neck, eyebrows, eyelashes, and vermilion were excluded from this calculation. The volar surface of 1 digit (the participant's thumb) was approximately 0.1% of the total body surface area and was used as a guide to estimate the baseline percentage of vitiligo involvement of face. The extent of depigmentation was expressed by the following percentages: 0, 10%, 25%, 50%, 75%, 90%, or 100%. Percent change from baseline in Local F-VASI = ((post baseline Local F-VASI - baseline Local F-VASI)/baseline Local F-VASI)×100. This outcome measure was the percentage of participants achieving at least 50% improvement in site assessment F-VASI from baseline (F-VASI50). Negative percent change from baseline in F-VASI signified an improvement. Baseline was defined as the last measurement prior to first dosing (Day 1).
Time Frame: Baseline, Weeks 4, 8, 12, 16, 20 and 24
Population: as for outcome 4
Measure: Number; unit: Percentage of Participants
Arm/Group | PF-06651600 200mg - 50mg QD | PF-06651600 100 mg - 50 mg QD | PF-06651600 50 mg QD | PF-06651600 30 mg QD | PF-06651600 10 mg QD | Placebo
Number analyzed (Participants) | 64 | 67 | 67 | 50 | 49 | 66
Percentage of Participants
  Week 4 | 3.1 | 3.0 | 1.5 | 2.0 | 0 | 3.0
  Week 8 | 9.4 | 3.0 | 4.5 | 2.0 | 4.1 | 4.5
  Week 12: number analyzed (Participants) | 62 | 66 | 66 | 49 | 48 | 66
  Week 12 | 16.1 | 9.1 | 9.1 | 8.2 | 8.3 | 9.1
  Week 16: number analyzed (Participants) | 63 | 62 | 66 | 47 | 47 | 63
  Week 16 | 14.3 | 9.7 | 13.6 | 8.5 | 10.6 | 14.3
  Week 20: number analyzed (Participants) | 61 | 67 | 64 | 49 | 48 | 63
  Week 20 | 18.0 | 14.9 | 17.2 | 12.2 | 16.7 | 17.5
  Week 24: number analyzed (Participants) | 63 | 65 | 65 | 47 | 49 | 66
  Week 24 | 20.6 | 21.5 | 15.4 | 10.6 | 18.4 | 16.7

18. Secondary Outcome: Percentage of Participants Achieving Local F-VASI75 at Designated Time Points - DR Period
Description: The site assessment of the F-VASI was calculated using a formula that included contribution from face (possible range, 0-4): Local F-VASI = [Digit Units] × [Depigmentation] × 0.1. Scalp, neck, eyebrows, eyelashes, and vermilion were excluded from this calculation. The volar surface of 1 digit (the participant's thumb) was approximately 0.1% of the total body surface area and was used as a guide to estimate the baseline percentage of vitiligo involvement of face. The extent of depigmentation was expressed by the following percentages: 0, 10%, 25%, 50%, 75%, 90%, or 100%. Percent change from baseline in Local F-VASI = ((post baseline Local F-VASI - baseline Local F-VASI)/baseline Local F-VASI)×100. This outcome measure was the percentage of participants achieving at least 75% improvement in site assessment F-VASI from baseline (F-VASI75). Negative percent change from baseline in F-VASI signified an improvement. Baseline was defined as the last measurement prior to first dosing (Day 1).
Time Frame: Baseline, Weeks 4, 8, 12, 16, 20 and 24
Population: as for outcome 4
Measure: Number; unit: Percentage of Participants
Arm/Group | PF-06651600 200mg - 50mg QD | PF-06651600 100 mg - 50 mg QD | PF-06651600 50 mg QD | PF-06651600 30 mg QD | PF-06651600 10 mg QD | Placebo
Number analyzed (Participants) | 64 | 67 | 67 | 50 | 49 | 66
Percentage of Participants
  Week 4 | 0 | 0 | 0 | 0 | 0 | 1.5
  Week 8 | 0 | 0 | 3.0 | 2.0 | 0 | 0
  Week 12: number analyzed (Participants) | 62 | 66 | 66 | 49 | 48 | 66
  Week 12 | 1.6 | 3.0 | 4.5 | 6.1 | 2.1 | 1.5
  Week 16: number analyzed (Participants) | 63 | 62 | 66 | 47 | 47 | 63
  Week 16 | 3.2 | 0 | 4.5 | 4.3 | 4.3 | 7.9
  Week 20: number analyzed (Participants) | 61 | 67 | 64 | 49 | 48 | 63
  Week 20 | 6.6 | 1.5 | 9.4 | 6.1 | 6.3 | 11.1
  Week 24: number analyzed (Participants) | 63 | 65 | 65 | 47 | 49 | 66
  Week 24 | 11.1 | 4.6 | 6.2 | 4.3 | 4.1 | 13.6

19. Secondary Outcome: Percentage of Participants Achieving Local F-VASI90 at Designated Time Points - DR Period
Description: The site assessment of the F-VASI was calculated using a formula that included contribution from face (possible range, 0-4): Local F-VASI = [Digit Units] × [Depigmentation] × 0.1. Scalp, neck, eyebrows, eyelashes, and vermilion were excluded from this calculation. The volar surface of 1 digit (the participant's thumb) was approximately 0.1% of the total body surface area and was used as a guide to estimate the baseline percentage of vitiligo involvement of face. The extent of depigmentation was expressed by the following percentages: 0, 10%, 25%, 50%, 75%, 90%, or 100%. Percent change from baseline in Local F-VASI = ((post baseline Local F-VASI - baseline Local F-VASI)/baseline Local F-VASI)×100. This outcome measure was the percentage of participants achieving at least 90% improvement in site assessment F-VASI from baseline (F-VASI90). Negative percent change from baseline in F-VASI signified an improvement. Baseline was defined as the last measurement prior to first dosing (Day 1).
Time Frame: Baseline, Weeks 4, 8, 12, 16, 20 and 24
Population: as for outcome 4
Measure: Number; unit: Percentage of Participants
Arm/Group | PF-06651600 200mg - 50mg QD | PF-06651600 100 mg - 50 mg QD | PF-06651600 50 mg QD | PF-06651600 30 mg QD | PF-06651600 10 mg QD | Placebo
Number analyzed (Participants) | 64 | 67 | 67 | 50 | 49 | 66
Percentage of Participants
  Week 4 | 0 | 0 | 0 | 0 | 0 | 0
  Week 8 | 0 | 0 | 1.5 | 2.0 | 0 | 0
  Week 12: number analyzed (Participants) | 62 | 66 | 66 | 49 | 48 | 66
  Week 12 | 0 | 0 | 1.5 | 2.0 | 0 | 0
  Week 16: number analyzed (Participants) | 63 | 62 | 66 | 47 | 47 | 63
  Week 16 | 1.6 | 0 | 3.0 | 2.1 | 2.1 | 0
  Week 20: number analyzed (Participants) | 61 | 67 | 64 | 49 | 48 | 63
  Week 20 | 1.6 | 1.5 | 4.7 | 2.0 | 2.1 | 1.6
  Week 24: number analyzed (Participants) | 63 | 65 | 65 | 47 | 49 | 66
  Week 24 | 1.6 | 1.5 | 3.1 | 0 | 4.1 | 1.5

20. Secondary Outcome: Percentage of Participants Achieving Local F-VASI100 at Designated Time Points - DR Period
Description: The site assessment of the F-VASI was calculated using a formula that included contribution from face (possible range, 0-4): Local F-VASI = [Digit Units] × [Depigmentation] × 0.1. Scalp, neck, eyebrows, eyelashes, and vermilion were excluded from this calculation. The volar surface of 1 digit (the participant's thumb) was approximately 0.1% of the total body surface area and was used as a guide to estimate the baseline percentage of vitiligo involvement of face. The extent of depigmentation was expressed by the following percentages: 0, 10%, 25%, 50%, 75%, 90%, or 100%. Percent change from baseline in Local F-VASI = ((post baseline Local F-VASI - baseline Local F-VASI)/baseline Local F-VASI)×100. This outcome measure was the percentage of participants achieving 100% improvement in site assessment F-VASI from baseline (F-VASI100). Negative percent change from baseline in F-VASI signified an improvement. Baseline was defined as the last measurement prior to first dosing (Day 1).
Time Frame: Baseline, Weeks 4, 8, 12, 16, 20 and 24
Population: as for outcome 4
Measure: Number; unit: Percentage of Participants
Arm/Group | PF-06651600 200mg - 50mg QD | PF-06651600 100 mg - 50 mg QD | PF-06651600 50 mg QD | PF-06651600 30 mg QD | PF-06651600 10 mg QD | Placebo
Number analyzed (Participants) | 64 | 67 | 67 | 50 | 49 | 66
Percentage of Participants
  Week 4 | 0 | 0 | 0 | 0 | 0 | 0
  Week 8 | 0 | 0 | 0 | 2.0 | 0 | 0
  Week 12: number analyzed (Participants) | 62 | 66 | 66 | 49 | 48 | 66
  Week 12 | 0 | 0 | 0 | 0 | 0 | 0
  Week 16: number analyzed (Participants) | 63 | 62 | 66 | 47 | 47 | 63
  Week 16 | 0 | 0 | 0 | 0 | 0 | 0
  Week 20: number analyzed (Participants) | 61 | 67 | 64 | 49 | 48 | 63
  Week 20 | 0 | 0 | 1.6 | 0 | 0 | 0
  Week 24: number analyzed (Participants) | 63 | 65 | 65 | 47 | 49 | 66
  Week 24 | 0 | 0 | 1.5 | 0 | 0 | 0

21. Secondary Outcome: Change From Baseline in Total VitiQoL Score at Designated Time Points - DR Period
Description: The Vitiligo-Specific Quality of Life (VitiQoL) instrument was a reliable and validated vitiligo disease-specific health-related quality of life (HRQoL) instrument which measured concepts relevant to vitiligo participants. The VitiQoL was a 15-item PRO measure which measured concepts of symptoms, daily activities, leisure activities, work, personal relationships and treatment. Responses ranged from "not at all" (scored 0) to "most of the time" (scored 6) and gave a minimum and maximum score from 0 to 90, with higher scores representing greater burden. The VitiQoL total score was calculated as sum of items 1-15.
  The change from baseline in total VitiQoL score was analyzed using the mixed-effect models repeated measures (MMRM) analysis. Baseline was defined as the last measurement prior to first dosing (Day 1).
Time Frame: Baseline, Weeks 4, 16 and 24
Population: as for outcome 4
Measure: Least Squares Mean (Standard Error); unit: Units on a Scale
Arm/Group | PF-06651600 200mg - 50mg QD | PF-06651600 100 mg - 50 mg QD | PF-06651600 50 mg QD | PF-06651600 30 mg QD | PF-06651600 10 mg QD | Placebo
Number analyzed (Participants) | 64 | 67 | 67 | 50 | 49 | 66
Units on a Scale
  Week 4: number analyzed (Participants) | 62 | 66 | 64 | 50 | 47 | 63
  Week 4 | -3.9 (1.34) | -2.9 (1.31) | -4.4 (1.31) | -4.4 (1.50) | -3.5 (1.54) | -5.1 (1.33)
  Week 16: number analyzed (Participants) | 54 | 56 | 56 | 41 | 44 | 59
  Week 16 | -6.5 (1.83) | -4.9 (1.79) | -6.3 (1.82) | -4.8 (2.07) | -10.5 (2.06) | -7.1 (1.78)
  Week 24: number analyzed (Participants) | 50 | 56 | 50 | 34 | 41 | 56
  Week 24 | -6.5 (1.99) | -3.6 (1.92) | -7.7 (1.99) | -7.0 (2.30) | -9.7 (2.22) | -6.4 (1.92)

22. Secondary Outcome: Change From Baseline in VitiQoL Participation Limitation Domain Score at Designated Time Points - DR Period
Description: The VitiQoL was a reliable and validated vitiligo disease specific HRQoL instrument which measured concepts relevant to vitiligo participants. The VitiQoL was a 15-item PRO measure which measured concepts of symptoms, daily activities, leisure activities, work, personal relationships and treatment. Responses ranged from "not at all" (scored 0) to "most of the time" (scored 6) and gave a minimum and maximum score from 0 to 90, with higher scores representing greater burden. The VitiQoL Participation Limitation domain score was the sum of items 3, 4, 6, 9, 10, 11, 14 and ranged from 0 to 42.
  The change from baseline in VitiQoL Participation Limitation Domain Score was analyzed using the MMRM analysis. Baseline was defined as the last measurement prior to first dosing (Day 1).
Time Frame: Baseline, Weeks 4, 16 and 24
Population: as for outcome 4
Measure: Least Squares Mean (Standard Error); unit: Units on a Scale
Arm/Group | PF-06651600 200mg - 50mg QD | PF-06651600 100 mg - 50 mg QD | PF-06651600 50 mg QD | PF-06651600 30 mg QD | PF-06651600 10 mg QD | Placebo
Number analyzed (Participants) | 64 | 67 | 67 | 50 | 49 | 66
Units on a Scale
  Week 4: number analyzed (Participants) | 62 | 66 | 64 | 50 | 47 | 63
  Week 4 | -1.2 (0.71) | -1.1 (0.69) | -1.7 (0.69) | -1.8 (0.79) | -1.0 (0.81) | -2.5 (0.70)
  Week 16: number analyzed (Participants) | 54 | 56 | 56 | 41 | 44 | 59
  Week 16 | -2.1 (0.88) | -1.9 (0.86) | -2.6 (0.87) | -2.3 (1.00) | -4.1 (0.99) | -3.1 (0.85)
  Week 24: number analyzed (Participants) | 50 | 56 | 50 | 34 | 41 | 56
  Week 24 | -1.4 (0.98) | -1.7 (0.94) | -3.2 (0.97) | -2.8 (1.14) | -3.9 (1.09) | -2.2 (0.94)

23. Secondary Outcome: Change From Baseline in VitiQoL Stigma Domain Score at Designated Time Points - DR Period
Description: The VitiQoL was a reliable and validated vitiligo disease specific HRQoL instrument which measured concepts relevant to vitiligo participants. The VitiQoL was a 15-item PRO measure which measured concepts of symptoms, daily activities, leisure activities, work, personal relationships and treatment. Responses ranged from "not at all" (scored 0) to "most of the time" (scored 6) and gave a minimum and maximum score from 0 to 90, with higher scores representing greater burden. The VitiQoL Stigma domain score was the sum of items 1, 2, 5, 7 and 15, and ranged from 0 to 30.
  The change from baseline in VitiQoL Stigma Domain Score was analyzed using the MMRM analysis. Baseline was defined as the last measurement prior to first dosing (Day 1).
Time Frame: Baseline, Weeks 4, 16 and 24
Population: as for outcome 4
Measure: Least Squares Mean (Standard Error); unit: Units on a Scale
Arm/Group | PF-06651600 200mg - 50mg QD | PF-06651600 100 mg - 50 mg QD | PF-06651600 50 mg QD | PF-06651600 30 mg QD | PF-06651600 10 mg QD | Placebo
Number analyzed (Participants) | 64 | 67 | 67 | 50 | 49 | 66
Units on a Scale
  Week 4: number analyzed (Participants) | 62 | 66 | 64 | 50 | 47 | 63
  Week 4 | -1.9 (0.56) | -1.6 (0.55) | -2.4 (0.55) | -1.7 (0.62) | -1.7 (0.64) | -1.8 (0.56)
  Week 16: number analyzed (Participants) | 54 | 56 | 56 | 41 | 44 | 59
  Week 16 | -3.4 (0.71) | -2.3 (0.70) | -3.2 (0.71) | -1.7 (0.80) | -4.3 (0.80) | -2.9 (0.69)
  Week 24: number analyzed (Participants) | 50 | 56 | 50 | 34 | 41 | 56
  Week 24 | -3.8 (0.76) | -2.1 (0.73) | -3.7 (0.76) | -3.1 (0.88) | -4.5 (0.84) | -3.2 (0.73)

24. Secondary Outcome: Change From Baseline in VitiQoL Behaviors Domain Score at Designated Time Points - DR Period
Description: The VitiQoL was a reliable and validated vitiligo disease specific HRQoL instrument which measured concepts relevant to vitiligo participants. The VitiQoL was a 15-item PRO measure which measured concepts of symptoms, daily activities, leisure activities, work, personal relationships and treatment. Responses ranged from "not at all" (scored 0) to "most of the time" (scored 6) and gave a minimum and maximum score from 0 to 90, with higher scores representing greater burden. The VitiQoL Behaviors domain score was the sum of items 8, 12 and 13, and ranged from 0 to 18.
  The change from baseline in VitiQoL Behaviors Domain Score was analyzed using the MMRM analysis. Baseline was defined as the last measurement prior to first dosing (Day 1).
Time Frame: Baseline, Weeks 4, 16 and 24
Population: as for outcome 4
Measure: Least Squares Mean (Standard Error); unit: Units on a Scale
Arm/Group | PF-06651600 200mg - 50mg QD | PF-06651600 100 mg - 50 mg QD | PF-06651600 50 mg QD | PF-06651600 30 mg QD | PF-06651600 10 mg QD | Placebo
Number analyzed (Participants) | 64 | 67 | 67 | 50 | 49 | 66
Units on a Scale
  Week 4: number analyzed (Participants) | 62 | 66 | 64 | 50 | 47 | 63
  Week 4 | -0.8 (0.37) | -0.3 (0.36) | -0.2 (0.36) | -0.9 (0.41) | -0.7 (0.42) | -0.7 (0.37)
  Week 16: number analyzed (Participants) | 54 | 56 | 56 | 41 | 44 | 59
  Week 16 | -1.1 (0.50) | -0.8 (0.49) | -0.5 (0.50) | -0.9 (0.57) | -2.1 (0.56) | -1.0 (0.49)
  Week 24: number analyzed (Participants) | 50 | 56 | 50 | 34 | 41 | 56
  Week 24 | -1.4 (0.53) | 0 (0.52) | -0.7 (0.53) | -1.3 (0.62) | -1.3 (0.60) | -0.9 (0.51)

25. Secondary Outcome: Percentage of Participants Achieving sIGA 0 or 1 and at Least a 2-Point Improvement at Week 24 - DR Period
Description: The percentage of participants achieving a static Investigator Global Assessment (sIGA) Score 0/1 and sIGA ≥2-point improvement at Week 24 was presented in this outcome measure. The sIGA score ranged from 0 to 4.
  The sIGA Score 0 represented "Clear" with no signs of loss of pigmentation with natural light or with Woods lamp examination.
  The sIGA Score 1 represented "Almost Clear" with the following descriptors:
  * Faint, barely detectable loss of pigmentation mainly located on dorsal hands, feet, bony prominences, and/or limited areas.
  * Approximately 90% pigmentation within lesions.
  * No or rare signs of Koebner phenomenon, confetti like or trichrome lesions could be present.
  The sIGA Scores 2, 3 and 4 represented "Mild Vitiligo", "Moderate Vitiligo" and "Severe Vitiligo", respectively.
Time Frame: Week 24
Population: as for outcome 1
Measure: Number; unit: Percentage of Participants
Arm/Group | PF-06651600 200mg - 50mg QD | PF-06651600 100 mg - 50 mg QD | PF-06651600 50 mg QD | PF-06651600 30 mg QD | PF-06651600 10 mg QD | Placebo
Number analyzed (Participants) | 62 | 64 | 65 | 46 | 48 | 65
Percentage of Participants | 0 | 0 | 0 | 0 | 0 | 0

26. Primary Outcome: Number of Participants With Treatment Emergent Adverse Events (TEAEs) and Serious Adverse Events (SAEs) up to Week 24 - DR Period
Description: Adverse Event (AE) was defined as any untoward medical occurrence in a study participant administered a product or medical device; the event did not necessarily need to have a causal relationship with the treatment or usage. An AE was considered a TEAE if the event started during the effective duration of treatment. All events that started on or after the first dosing day and time/start time, if collected, but before the last dose plus the lag time were flagged as TEAEs. SAE was defined as any untoward medical occurrence at any dose that resulted in death; was life threatening (immediate risk of death); required inpatient hospitalization or prolongation of existing hospitalization; resulted in persistent or significant disability/incapacity (substantial disruption of the ability to conduct normal life functions); resulted in congenital anomaly/birth defect; or that was considered to be an important medical event. Causality to study treatment was determined by the investigator.
Time Frame: 24 weeks
Population: The safety analysis population included all participants who received at least 1 dose of investigational product.
Measure: Count of Participants; unit: Participants
Arm/Group | PF-06651600 200 mg - 50 mg QD | PF-06651600 100 mg - 50 mg QD | PF-06651600 50 mg QD | PF-06651600 30 mg QD | PF-06651600 10 mg QD | Placebo
Number analyzed (Participants) | 65 | 67 | 67 | 50 | 49 | 66
Participants
  Participants With All-Causality TEAEs | 56 | 45 | 54 | 30 | 40 | 52
  Participants With Treatment-Related TEAEs | 32 | 19 | 20 | 17 | 18 | 20
  Participants With All-Causality SAEs | 0 | 0 | 1 | 1 | 1 | 1
  Participants With Treatment-Related SAEs | 0 | 0 | 0 | 0 | 0 | 0

27. Primary Outcome: Number of Participants With the TEAEs of Anaemia, Neutropenia, Thrombocytopenia and Lymphopenia - DR Period
Description: An AE was any untoward medical occurrence in a study participant administered a product or medical device; the event did not necessarily need to have a causal relationship with the treatment or usage. The abnormal test findings, clinically significant signs and symptoms of anaemia, neutropenia, thrombocytopenia and lymphopenia were reported as AEs. The clinical significance was determined by the investigator.
  An AE was considered a TEAE if the event started during the effective duration of treatment. All events that started on or after the first dosing day and time/start time, if collected, but before the last dose plus the lag time were flagged as TEAEs.
  Baseline was defined as the last measurement prior to first dosing (Day 1).
Time Frame: Baseline up to Week 24
Population: The safety analysis population included all participants who received at least 1 dose of investigational product.
Measure: Count of Participants; unit: Participants
Arm/Group | PF-06651600 200mg - 50mg QD | PF-06651600 100 mg - 50 mg QD | PF-06651600 50 mg QD | PF-06651600 30 mg QD | PF-06651600 10 mg QD | Placebo
Number analyzed (Participants) | 65 | 67 | 67 | 50 | 49 | 66
Participants
  Participants With Anaemia | 0 | 0 | 0 | 0 | 0 | 0
  Participants With Neutropenia | 0 | 1 | 0 | 0 | 1 | 1
  Participants With Thrombocytopenia | 1 | 0 | 0 | 0 | 0 | 0
  Participants With Lymphopenia | 1 | 0 | 0 | 0 | 0 | 0

28. Primary Outcome: Number of Participants With Clinically Meaningful Changes From Baseline in Lipid Profile up to Week 24 - DR Period
Description: Participants had to abstain from all food and drink (except water and non-investigational products) for an 8-hour overnight fast prior to fasting lipid profile panel collection. Fasting lipid assessment included total cholesterol, low-density lipoprotein (LDL) cholesterol, high-density lipoprotein (HDL) cholesterol, and triglycerides. The clinical meaningfulness was determined by the investigator.
  Baseline was defined as the last measurement prior to first dosing (Day 1).
Time Frame: Baseline up to Week 24
Population: The safety analysis population included all participants who received at least 1 dose of investigational product.
Measure: Count of Participants; unit: Participants
Arm/Group | PF-06651600 200 mg - 50 mg QD | PF-06651600 100 mg - 50 mg QD | PF-06651600 50 mg QD | PF-06651600 30 mg QD | PF-06651600 10 mg QD | Placebo
Number analyzed (Participants) | 65 | 67 | 67 | 50 | 49 | 66
Participants | 0 | 0 | 0 | 0 | 0 | 0

29. Primary Outcome: Number of Participants With Liver Function Test Values Meeting the Protocol-Specified Discontinuation Criteria - DR Period
Description: Liver function tests included tests of alanine aminotransferase (ALT), aspartate aminotransferase (AST) and total bilirubin.
Time Frame: 24 weeks
Population: The safety analysis population included all participants who received at least 1 dose of investigational product.
Measure: Count of Participants; unit: Participants
Arm/Group | PF-06651600 200 mg - 50 mg QD | PF-06651600 100 mg - 50 mg QD | PF-06651600 50 mg QD | PF-06651600 30 mg QD | PF-06651600 10 mg QD | Placebo
Number analyzed (Participants) | 65 | 67 | 67 | 50 | 49 | 66
Participants
  Bilirubin > 1.5 x upper limit of normal (ULN) | 0 | 0 | 0 | 0 | 0 | 0
  AST > 2.5 x ULN | 1 | 0 | 1 | 0 | 1 | 0
  ALT > 2.5 x ULN | 0 | 0 | 1 | 1 | 1 | 1

30. Primary Outcome: Number of Participants With TEAEs and SAEs - Extension (Ext) Period
Description: AE was defined as any untoward medical occurrence in a study participant administered a product or medical device; the event did not necessarily need to have a causal relationship with the treatment or usage. An AE was considered a TEAE if the event started during the effective duration of treatment. All events that started on or after the first dosing day and time/start time, if collected, but before the last dose plus the lag time were flagged as TEAEs. SAE was defined as any untoward medical occurrence at any dose that resulted in death; was life threatening (immediate risk of death); requires inpatient hospitalization or prolongation of existing hospitalization; resulted in persistent or significant disability/incapacity (substantial disruption of the ability to conduct normal life functions); resulted in congenital anomaly/birth defect; or that was considered to be an important medical event. Causality to study treatment was determined by the investigator.
Time Frame: 24 weeks
Population: The safety analysis population included all participants who received at least 1 dose of investigational product.
Measure: Count of Participants; unit: Participants
Arm/Group | Extension (EXT) PF-06700841 60 mg - 30 mg QD | EXT PF-06651600 200 Mg-50 mg QD + nbUVB | EXT PF-06651600 200 mg - 50 mg QD | EXT PF-06651600 50 mg QD | EXT PF-06651600 30 mg QD
Number analyzed (Participants) | 55 | 43 | 187 | 6 | 2
Participants
  Participants With All-Causality TEAEs | 38 | 32 | 119 | 3 | 2
  Participants With Treatment-Related TEAEs | 20 | 12 | 36 | 0 | 0
  Participants With All-Causality SAEs | 1 | 0 | 1 | 0 | 0
  Participants With Treatment-Related SAEs | 1 | 0 | 0 | 0 | 0

31. Primary Outcome: Number of Participants With the TEAEs of Anaemia, Neutropenia, Thrombocytopenia and Lymphopenia - Ext Period
Description: An AE was any untoward medical occurrence in a study participant administered a product or medical device; the event did not necessarily need to have a causal relationship with the treatment or usage. The abnormal test findings, clinically significant signs and symptoms of anaemia, neutropenia, thrombocytopenia and lymphopenia were reported as AEs. The clinical significance was determined by the investigator.
  An AE was considered a TEAE if the event started during the effective duration of treatment. All events that started on or after the first dosing day and time/start time, if collected, but before the last dose plus the lag time were flagged as TEAEs.
Time Frame: 24 weeks
Population: The safety analysis population included all participants who received at least 1 dose of investigational product.
Measure: Count of Participants; unit: Participants
Groups:
- EX PF-06651600 50mg QD: 50 mg QD of PF 06651600 for 24 weeks. This arm is double blinded.
Arm/Group | Extension (EXT) PF-06700841 60 mg - 30 mg QD | EXT PF-06651600 200 Mg-50 mg QD + nbUVB | EXT PF-06651600 200 mg - 50 mg QD | EX PF-06651600 50mg QD | EXT PF-06651600 30 mg QD
Number analyzed (Participants) | 55 | 43 | 187 | 6 | 2
Participants
  Participants With Anemia | 0 | 0 | 0 | 1 | 0
  Participants With Neutropenia | 1 | 0 | 1 | 0 | 0
  Participants With Thrombocytopenia | 0 | 0 | 0 | 0 | 0
  Participants With Lymphopenia | 0 | 0 | 0 | 0 | 0

32. Primary Outcome: Number of Participants With Clinically Meaningful Changes From Baseline in Lipid Profile - Ext Period
Description: Participants had to abstain from all food and drink (except water and non-investigational products) for an 8-hour overnight fast prior to fasting lipid profile panel collection. Fasting lipid assessment included total cholesterol, LDL cholesterol, HDL cholesterol, and triglycerides. The clinical meaningfulness was determined by the investigator.
Time Frame: 24 Weeks
Population: The safety analysis population included all participants who received at least 1 dose of investigational product.
Measure: Count of Participants; unit: Participants
Arm/Group | Extension (EXT) PF-06700841 60 mg - 30 mg QD | EXT PF-06651600 200 Mg-50 mg QD + nbUVB | EXT PF-06651600 200 mg - 50 mg QD | EXT PF-06651600 50 mg QD | EXT PF-06651600 30 mg QD
Number analyzed (Participants) | 55 | 43 | 187 | 6 | 2
Participants | 0 | 0 | 0 | 0 | 0

33. Primary Outcome: Number of Participants With Liver Function Test Values Meeting the Protocol-Specified Discontinuation Criteria - Ext Period
Description: as for outcome 29
Time Frame: 24 weeks
Population: The safety analysis population included all participants who received at least 1 dose of investigational product. Number of participants analyzed signifies number of participants who were evaluable for this outcome measure.
Measure: Count of Participants; unit: Participants
Arm/Group | Extension (EXT) PF-06700841 60 mg - 30 mg QD | EXT PF-06651600 200 Mg-50 mg QD + nbUVB | EXT PF-06651600 200 mg - 50 mg QD | EXT PF-06651600 50 mg QD | EXT PF-06651600 30 mg QD
Number analyzed (Participants) | 55 | 42 | 186 | 6 | 2
Participants
  Bilirubin > 1.5 x ULN | 0 | 0 | 0 | 0 | 0
  AST > 2.5 x ULN | 0 | 0 | 0 | 0 | 0
  ALT > 2.5 x ULN | 0 | 0 | 1 | 0 | 0

ADVERSE EVENTS:
Time Frame: 48 weeks
Description: The same event may appear as both an AE and a SAE. However, what is presented are distinct events. An event may be categorized as serious in one participant and as non-serious in another participant, or one participant may have experienced both a serious and non-serious event during the study.
Groups:
- EX PF-06651600 200 mg - 50 mg QD + nbUVB: Induction dose of PF-06651600 200 mg QD plus standardized narrow band UVB (nbUVB) add-on therapy for 4 weeks followed by maintenance dosing of PF-06651600 50 mg QD plus standardized nbUVB add-on therapy for 20 weeks (only for participants who provide nbUVB consent). Participants who had <10% improvement in percent change in VASI at Extension Week 12 from the baseline value at Dose Ranging Period Week 24 were discontinued from the treatment and entered Follow-up Period. This arm is open label.
- EX PF-06651600 200mg-50mg QD: Induction dose of 200 mg QD of PF 06651600 for 4 weeks followed by maintenance dosing of 50 mg QD of PF 06651600 for 20 weeks. This arm is double blinded.
Arm/Group | PF-06651600 200 mg - 50 mg QD | PF-06651600 100 mg - 50 mg QD | PF-06651600 50 mg QD | PF-06651600 30 mg QD | PF-06651600 10 mg QD | Placebo | Extension (EXT) PF-06700841 60 mg - 30 mg QD | EX PF-06651600 200 mg - 50 mg QD + nbUVB | EX PF-06651600 200mg-50mg QD | EX PF-06651600 50mg QD | EXT PF-06651600 30 mg QD
All-Cause Mortality (participants affected / at risk) | 0/65 | 0/67 | 0/67 | 0/50 | 0/49 | 0/66 | 0/55 | 0/43 | 0/187 | 0/6 | 0/2
Serious Adverse Events (participants affected / at risk) | 0/65 | 0/67 | 1/67 | 1/50 | 1/49 | 1/66 | 1/55 | 0/43 | 1/187 | 0/6 | 0/2
Other Adverse Events (participants affected / at risk) | 31/65 | 35/67 | 32/67 | 23/50 | 22/49 | 37/66 | 17/55 | 14/43 | 46/187 | 3/6 | 2/2
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | PF-06651600 200 mg - 50 mg QD (N=65) | PF-06651600 100 mg - 50 mg QD (N=67) | PF-06651600 50 mg QD (N=67) | PF-06651600 30 mg QD (N=50) | PF-06651600 10 mg QD (N=49) | Placebo (N=66) | Extension (EXT) PF-06700841 60 mg - 30 mg QD (N=55) | EX PF-06651600 200 mg - 50 mg QD + nbUVB (N=43) | EX PF-06651600 200mg-50mg QD (N=187) | EX PF-06651600 50mg QD (N=6) | EXT PF-06651600 30 mg QD (N=2)
Oesophageal spasm (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Migraine (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Neurogenic bladder (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Disseminated varicella zoster virus infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Uterine leiomyoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | PF-06651600 200 mg - 50 mg QD (N=65) | PF-06651600 100 mg - 50 mg QD (N=67) | PF-06651600 50 mg QD (N=67) | PF-06651600 30 mg QD (N=50) | PF-06651600 10 mg QD (N=49) | Placebo (N=66) | Extension (EXT) PF-06700841 60 mg - 30 mg QD (N=55) | EX PF-06651600 200 mg - 50 mg QD + nbUVB (N=43) | EX PF-06651600 200mg-50mg QD (N=187) | EX PF-06651600 50mg QD (N=6) | EXT PF-06651600 30 mg QD (N=2)
Abdominal pain (Gastrointestinal disorders) | 0 (0) | 1 (1) | 2 (3) | 0 (0) | 1 (1) | 4 (4) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Diarrhoea (Gastrointestinal disorders) | 0 (0) | 5 (7) | 2 (2) | 4 (5) | 1 (1) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Dyspepsia (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 3 (4) | 3 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Fatigue (General disorders) | 6 (6) | 1 (1) | 2 (2) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Bronchitis (Infections and infestations) | 0 (0) | 1 (1) | 1 (1) | 3 (6) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Folliculitis (Infections and infestations) | 0 (0) | 1 (2) | 1 (1) | 1 (1) | 0 (0) | 4 (4) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Gastroenteritis (Infections and infestations) | 2 (2) | 0 (0) | 1 (1) | 3 (3) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Nasopharyngitis (Infections and infestations) | 8 (9) | 10 (11) | 16 (20) | 5 (8) | 5 (5) | 14 (20) | 3 (3) | 0 (0) | 8 (10) | 0 (0) | 0 (0)
Upper respiratory tract infection (Infections and infestations) | 5 (6) | 10 (11) | 5 (8) | 8 (8) | 6 (7) | 8 (8) | 4 (4) | 2 (2) | 9 (10) | 0 (0) | 0 (0)
Urinary tract infection (Infections and infestations) | 4 (5) | 4 (6) | 2 (2) | 2 (2) | 3 (3) | 3 (3) | 1 (2) | 3 (4) | 12 (16) | 1 (1) | 1 (1)
Back pain (Musculoskeletal and connective tissue disorders) | 3 (3) | 3 (3) | 6 (8) | 0 (0) | 1 (1) | 3 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Headache (Nervous system disorders) | 4 (4) | 7 (9) | 8 (8) | 1 (2) | 4 (5) | 8 (10) | 4 (4) | 3 (3) | 8 (8) | 0 (0) | 0 (0)
Acne (Skin and subcutaneous tissue disorders) | 4 (4) | 1 (1) | 4 (4) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Dry skin (Skin and subcutaneous tissue disorders) | 1 (1) | 4 (4) | 0 (0) | 2 (2) | 1 (1) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pruritus (Skin and subcutaneous tissue disorders) | 3 (3) | 2 (2) | 2 (2) | 1 (1) | 2 (2) | 5 (5) | 0 (0) | 3 (3) | 5 (6) | 0 (0) | 0 (0)
Urticaria (Skin and subcutaneous tissue disorders) | 2 (3) | 3 (6) | 1 (1) | 0 (0) | 3 (4) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Anaemia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Ear pain (Ear and labyrinth disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Influenza like illness (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
COVID-19 (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 1 (1)
Influenza (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 3 (3) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Onychomycosis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Blood creatine phosphokinase increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 3 (3) | 4 (5) | 3 (3) | 0 (0) | 0 (0)
Hypercholesterolaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Spinal segmental dysfunction (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Cough (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 3 (3) | 2 (2) | 3 (3) | 0 (0) | 0 (0)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Photosensitivity reaction (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 3 (4) | 0 (0) | 0 (0) | 0 (0)
Rash (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (3) | 0 (0) | 1 (1)
Hypertension (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 2 (2) | 1 (1) | 0 (0)
Insomnia (Psychiatric disorders) | 1 (1) | 0 (0) | 1 (1) | 3 (3) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Pfizer has the right to review disclosures, requesting a delay of less than 60 days. Investigator will postpone single center publications until after disclosure of pooled data (all sites), less than 12 months from study completion/termination at all participating sites. Investigator may not disclose previously undisclosed confidential information other than study results.

DOCUMENTS (2):
  • Study Protocol (2020-06-26): https://cdn.clinicaltrials.gov/large-docs/29/NCT03715829/Prot_000.pdf
  • Statistical Analysis Plan (2021-02-25): https://cdn.clinicaltrials.gov/large-docs/29/NCT03715829/SAP_001.pdf